CLINICAL TRIAL: NCT01631825
Title: An Open-label Long-term Extension Trial From Phase III of SPM962 (243-08-002) in Advanced Parkinson's Disease Patients With Concomitant Treatment of L-dopa
Brief Title: A Long-Term Extension Trial From of SPM 962 in Advanced Parkinson's Disease Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 243-08-002
Record Dates: First submitted 2012-06-25; First posted 2012-06-29 (Estimated); Results first posted 2014-03-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-02

CONDITIONS: Parkinson's Disease
Keywords: SPM 962; rotigotine; Parkinson's disease; concomitant use of L-dopa
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SPM 962 (Experimental): SPM 962 transdermal patch
  Interventions: Drug: SPM 962

INTERVENTIONS:
Drug: SPM 962 — SPM 962 transdermal patch once a daily up to 36.0 mg/day
  Other Names: rotigotine

SUMMARY:
* To investigate the safety of once-daily repeated transdermal administration of SPM 962 within a dose range of 4.5 to 36.0 mg/day (54-week treatment period) in Parkinson's disease (PD) patients treated concomitantly with L-dopa in a multi-center, open-label uncontrolled study.
* To investigate efficacy of SPM 962 in an exploratory manner.

ELIGIBILITY:
Inclusion Criteria:

* Subject completed the preceding trial 243-08-001.

Exclusion Criteria:

* Subject discontinued from the preceding trial 243-08-001.
* Subject had a serious adverse event which association with the investigational drug was not ruled out during trial 243-08-001.
* Subject has a persistent serious adverse event at the baseline, which was observed and association with the investigational drug was ruled out during trial 243-08-001.
* Subject had persistent confusion, hallucination, delusion or excitation during trial 243-08-001.
* Subject has abnormal behavior such as obsessive-compulsive disorder and delusion in 243-08-001 study.
* Subject showed serious or extensive application site reactions beyond the application site in the 243-08-001 study.
* Subject has orthostatic hypotension or a systolic blood pressure (SBP) <= 100 mmHg and has a decrease of SBP from spine to standing position >= 30 mmHg at baseline.
* Subject has a history of epilepsy, convulsion etc. during trial 243-08-001.
* Subject develops serious ECG abnormality at the baseline.
* Subject has QTc-interval >= 500 msec at the baseline or subject has an increase of QTc-interval >= 60 msec from the baseline in the trial 243-08-001 and has a QTc-interval > 470 msec in female or > 450 msec in male at the baseline.
* Subject had a serum potassium level < 3.5 mEq/L at the end of the taper period in trial 243-08-001.
* Subject has a total bilirubin >= 3.0 mg/dL or AST(GOT) or ALT(GPT) greater than 2.5 times of the upper limit of the reference range (or ? 100 IU/L) at the end of the period in trial 243-08-001.
* Subject had BUN >= 30 mg/dL or serum creatinine >= 2.0 mg/dl at the end of the taper period in trial 243-08-001.
* Subject who plans pregnancy during the trial.
* Subject is unable to give consent.
* Subject is judged to be inappropriate for this trial by the investigator for the reasons other than above.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2009-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyoji Imaoka, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (8):
- Japan (8):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SPM 962
Started | 321
Completed | 256
Not Completed | 65
Not completed — Adverse Event | 42
Not completed — Lack of Efficacy | 7
Not completed — Withdrawal by Subject | 9
Not completed — Protocol Violation | 4
Not completed — Discontinuation criteria | 1
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | SPM 962
Number analyzed (Participants) | 321
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (8.4)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 115
  >=65 years | 206
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 185
  Male | 136
Region of Enrollment [Number; unit: participants]
  Japan | 321

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Adverse Events (AEs), Vital Signs, and Laboratory Parameters
Description: The safety of the long-term SPM 962 treatment was examined based on the incidence and severity of AEs, vital signs, and laboratory parameters.
  AEs of special interest (1-3) are defined as below:
  1. sudden onset of sleep
  2. obsessive-compulsive disorder or impulse-control disorder
  3. hallucination, delusion
  Application site reaction is scored as -, ±, +, ++, +++, or ++++. More + indicates a greater severity of symptoms. The worst score obtained throughout the evaluation period was to be assessed.
Time Frame: Up to 55 weeks after dosing
Population: Safety set (SS)
Measure: Number; unit: participants
Arm/Group | SPM 962
Number analyzed (Participants) | 321
participants
  Any AEs | 311
  Treatment-related AEs | 269
  SAEs | 34
  Treatment-related SAEs | 6
  Severe AEs | 16
  Discontinuation due to AEs | 47
  Death | 1
  AEs of special interest 1 | 7
  AEs of special interest 2 | 4
  AEs of special interest 3 | 54
  Valvular disease of the heart | 0
  Sitting systolic blood pressure, ≤ 100 mmHg | 9
  QTcB ≥ 500 ms | 5
  QTcF ≥ 500 ms | 2
  Application site reaction ≥ +++ | 14
  Weight decrease reported as AE | 8

2. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Part 3 Sum Score
Description: Mean change (LOCF) from baseline in UPDRS Part 3 sum score (on state).
  UPDRS is a scale for monitoring Parkinson's Disease-related disability and impairment. The UPDRS consists of the following four sub-scales. Part 1: Mentation, Part 2: Activities of Daily Living, Part 3: Motor, Part 4: Complications. Part 3 assesses 14 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, Up to 54 weeks after dosing
Population: Full analysis set (FAS), last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962
Number analyzed (Participants) | 316
Scores on a scale
  Week 12 | -8.3 (7.1)
  Week 24 | -8.0 (7.6)
  Week 52 | -7.5 (8.6)

3. Secondary Outcome: UPDRS Part 2 Sum Score (Average of on State and Off State)
Description: Mean change (LOCF) from baseline in UPDRS Part 2 sum score (average of on state and off state).
  UPDRS sub-scale Part 2 assesses 13 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, up to 54 weeks after dosing
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962
Number analyzed (Participants) | 316
Scores on a scale
  Week 12 | -2.6 (3.0)
  Week 24 | -2.5 (3.4)
  Week 52 | -1.9 (4.0)

4. Secondary Outcome: Absolute Time Spent "Off"
Description: Mean number of hours in "off state" during a 24-hour period.
Time Frame: Baseline, up to 54 weeks after dosing
Population: FAS subjects with measurable off time at baseline, LOCF
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | SPM 962
Number analyzed (Participants) | 213
Hours
  Week 12 | -2.5 (2.5)
  Week 24 | -2.5 (2.7)
  Week 52 | -2.0 (2.7)

5. Secondary Outcome: UPDRS Part 1 Sum Score
Description: Mean change (LOCF) from baseline in UPDRS Part 1 sum score.
  UPDRS sub-scale Part 1 assesses 4 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, up to 54 weeks after dosing
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962
Number analyzed (Participants) | 317
Scores on a scale
  Week 12 | -0.33 (1.07)
  Week 24 | -0.25 (1.17)
  Week 52 | -0.15 (1.29)

6. Secondary Outcome: UPDRS Part 2 Sum Score (On State)
Description: Mean change (LOCF) from baseline in UPDRS Part 2 sum score (on state). A decrease in the scores means improvement.
Time Frame: Baseline, up to 54 weeks after dosing
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962
Number analyzed (Participants) | 317
Scores on a scale
  Week 12 | -1.9 (2.8)
  Week 24 | -1.7 (3.0)
  Week 52 | -1.3 (3.7)

7. Secondary Outcome: UPDRS Part 2 Sum Score (Off State)
Description: Mean change (LOCF) from baseline in UPDRS Part 2 sum score (off state). A decrease in the scores means improvement.
Time Frame: Baseline, up to 54 weeks after dosing
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962
Number analyzed (Participants) | 212
Scores on a scale
  Week 12 | -3.7 (4.3)
  Week 24 | -3.8 (4.8)
  Week 52 | -2.5 (5.5)

8. Secondary Outcome: UPDRS Part 4 Sum Score
Description: Mean change (LOCF) from baseline in UPDRS Part 4 sum score.
  UPDRS sub-scale Part 4 assesses 11 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score.
  A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, up to 54 weeks after dosing
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962
Number analyzed (Participants) | 317
Scores on a scale
  Week 12 | -0.24 (1.29)
  Week 24 | -0.28 (1.32)
  Week 52 | -0.13 (1.42)

9. Secondary Outcome: Total of UPDRS Part 1 Sum Score, UPDRS Part 2 Sum Score (Average of on State and Off State), UPDRS Part 3 Sum Score (on State), and UPDRS Part 4 Sum Score
Description: Mean change (LOCF) from baseline in total of UPDRS Part 1 sum score, UPDRS Part 2 sum score (average of on state and off state), UPDRS Part 3 sum score (on state), and UPDRS Part 4 sum score.
  A decrease in the scores means improvement.
Time Frame: Baseline, up to 54 weeks after dosing
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962
Number analyzed (Participants) | 315
Scores on a scale
  Week 12 | -11.4 (9.7)
  Week 24 | -11.1 (10.5)
  Week 52 | -9.7 (12.1)

10. Secondary Outcome: The Modified Hoehn & Yahr Severity of Illness
Description: Change (LOCF) from baseline in the Modified Hoehn & Yahr Severity of Illness. The Modified Hoehn & Yahr criteria are measured on the following 8-point scale for staging: 0, No signs of disease; 1, Unilateral disease; 1.5, Unilateral plus axial involvement; 2, Bilateral disease without impairment of balance; 2.5, Mild bilateral disease with recovery on pull test; 3, Mild to moderate bilateral disease, some postural instability, physically independent 4, Severe disability, still able to walk or stand unassisted; and 5, Wheelchair bound or bedridden unless aided.
  The data at week 52 is shown.
Time Frame: Baseline, up to 54 weeks after dosing.
Population: FAS, LOCF
Measure: Number; unit: Percentage of participants
Arm/Group | SPM 962
Number analyzed (Participants) | 316
Percentage of participants
  Increased | 7.3
  Not changed | 62.5
  Decreased | 30.2

11. Secondary Outcome: Each Item of UPDRS Part 1
Description: The percentage of subjects with elevated scores for each item of UPDRS Part 1. The data at week 52 is shown.
Time Frame: Baseline, up to 54 weeks after dosing.
Population: FAS, LOCF
Measure: Number; unit: Percentage of Participants
Arm/Group | SPM 962
Number analyzed (Participants) | 317
Percentage of Participants
  Intellectual impairment | 2.8
  Thought disorder | 9.5
  Depression | 5.0
  Motivation/Initiative | 4.4

12. Secondary Outcome: Each Item of UPDRS Part 2 (on State)
Description: The percentage of subjects with elevated scores for each item of UPDRS Part 2 (on state). The data at week 52 is shown.
Time Frame: Baseline, up to 54 weeks after dosing.
Population: FAS, LOCF
Measure: Number; unit: Percentage of Participants
Arm/Group | SPM 962
Number analyzed (Participants) | 317
Percentage of Participants
  Speech | 4.7
  Salivation | 11.0
  Swallowing | 6.0
  Handwriting | 7.6
  Cutting Food and Handling Utensils | 6.9
  Dressing | 6.6
  Hygiene | 5.0
  Turning in Bed / Adjusting Bed Clothes | 7.9
  Falling - Unrelated to Freezing | 8.2
  Freezing When Walking | 6.6
  Walking | 8.5
  Tremor | 4.4
  Sensory Complaints Related to Parkinsonism | 3.5

13. Secondary Outcome: Each Item of UPDRS Part 2 (Off State)
Description: The percentage of subjects with elevated scores for each item of UPDRS Part 2 (off state). The data at week 52 is shown.
Time Frame: Baseline, up to 54 weeks after dosing.
Population: FAS, LOCF
Measure: Number; unit: Percentage of Participants
Arm/Group | SPM 962
Number analyzed (Participants) | 190
Percentage of Participants
  Speech | 5.8
  Salivation | 10.5
  Swallowing | 6.3
  Handwriting | 11.6
  Cutting Food and Handling Utensils | 11.6
  Dressing | 9.5
  Hygiene | 11.6
  Turning in Bed / Adjusting Bed Clothes | 10.5
  Falling - Unrelated to Freezing | 9.5
  Freezing When Walking | 17.9
  Walking | 13.2
  Tremor | 4.2
  Sensory Complaints Related to Parkinsonism | 5.8

14. Secondary Outcome: Each Item of UPDRS Part 2 (Average of on State and Off State)
Description: The percentage of subjects with elevated scores for each item of UPDRS Part 2 (average of on state and off state). The data at week 52 is shown.
Time Frame: Baseline, up to 54 weeks after dosing.
Population: FAS, LOCF
Measure: Number; unit: Percentage of Participants
Arm/Group | SPM 962
Number analyzed (Participants) | 317
Percentage of Participants
  Speech | 6.7
  Salivation | 13.7
  Swallowing | 7.6
  Handwriting | 12.1
  Cutting Food and Handling Utensils | 11.1
  Dressing | 9.2
  Hygiene | 10.2
  Turning in Bed / Adjusting Bed Clothes | 10.5
  Falling - Unrelated to Freezing | 9.9
  Freezing When Walking | 14.6
  Walking | 12.7
  Tremor | 5.7
  Sensory Complaints Related to Parkinsonism | 5.7

15. Secondary Outcome: Total of UPDRS Part 2 Sum Score (Average of on State and Off State) and UPDRS Part 3 Sum Score (on State)
Description: Mean change (LOCF) from baseline in total of UPDRS Part 2 sum score (average of on state and off state) and UPDRS Part 3 sum score (on state).
  A decrease in the scores means improvement.
Time Frame: Baseline, up to 54 weeks after dosing
Population: FAS, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962
Number analyzed (Participants) | 315
Scores on a scale
  Week 12 | -10.9 (9.2)
  Week 24 | -10.5 (9.9)
  Week 52 | -9.4 (11.4)

16. Secondary Outcome: Each Item of UPDRS Part 3 (on State)
Description: The percentage of subjects with elevated scores for each item of UPDRS Part 3 (on state). The data at week 52 is shown.
Time Frame: Baseline, up to 54 weeks after dosing.
Population: FAS, LOCF
Measure: Number; unit: Percentage of Participants
Arm/Group | SPM 962
Number analyzed (Participants) | 317
Percentage of Participants
  Speech | 6.3
  Facial Expression | 5.4
  Tremor at Rest (Face, lips, chin) | 0.6
  Tremor at Rest (Left hand) | 1.6
  Tremor at Rest (Right hand) | 1.6
  Tremor at Rest (Left foot) | 2.2
  Tremor at Rest (Right foot) | 1.6
  Action or Postural Tremor of Hands (Left hand) | 5.4
  Action or Postural Tremor of Hands (Right hand) | 6.6
  Rigidity (Neck) | 5.0
  Rigidity (Left upper extremity) | 2.8
  Rigidity (Right upper extremity) | 2.8
  Rigidity (Left lower extremity) | 5.0
  Rigidity (Right lower extremity) | 4.1
  Finger Taps (Left) | 5.1
  Finger Taps (Right) | 5.7
  Hand Movements (Left) | 7.6
  Hand Movements (Right) | 6.6
  Rapid Alternating Movements of Hands (Left) | 7.3
  Rapid Alternating Movements of Hands (Right) | 6.9
  Leg Agility (Left) | 6.6
  Leg Agility (Right) | 7.3
  Arising From Chair | 9.6
  Posture Erect | 11.4
  Gait | 9.6
  Postural Stability | 8.9
  Body Bradykinesia / Hypokinesia | 7.0

17. Secondary Outcome: Each Item of UPDRS Part 4
Description: The percentage of subjects with elevated scores for each item of UPDRS Part 4. The data at week 52 is shown.
Time Frame: Baseline, up to 54 weeks after dosing.
Population: FAS, LOCF
Measure: Number; unit: Percentage of Participants
Arm/Group | SPM 962
Number analyzed (Participants) | 317
Percentage of Participants
  Duration | 15.1
  Disability | 5.7
  Painful Dyskinesias | 0.6
  Presence of Early Morning Dystonia | 2.5
  Are "off" periods predictable? | 3.2
  Are "off" periods unpredictable? | 1.6
  Do "off" periods come on suddenly? | 1.3
  Proportion of "off" in waking day | 5.7
  Patients with anorexia, nausea, or vomiting | 5.0
  Patients with any sleep disturbances | 10.7
  Patient with symptomatic orthostasis | 1.9

ADVERSE EVENTS:
Time Frame: 54 weeks
Arm/Group | SPM 962
Serious Adverse Events (participants affected / at risk) | 34/321
Other Adverse Events (participants affected / at risk) | 290/321
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPM 962 (N=321)
Colonic Polyp (Gastrointestinal disorders) | 1 (1)
Gastric Ulcer Bleeding (Gastrointestinal disorders) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Hernia Inguinal (Gastrointestinal disorders) | 1 (1)
Sudden Death (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Septicaemia (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1)
Haematoma Subdural (Injury, poisoning and procedural complications) | 2 (2)
Heat Illness (Injury, poisoning and procedural complications) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1)
Jaw Fracture (Injury, poisoning and procedural complications) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 (1)
Ulna Fracture (Injury, poisoning and procedural complications) | 1 (1)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Extranodal Marginal Zone B-Cell Lymphoma (Malt Type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Large Intestine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carpal Tunnel Syndrome (Nervous system disorders) | 1 (1)
Depressed Level Of Consciousness (Nervous system disorders) | 2 (2)
Disease Parkinson's (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Hallucination Visual (Psychiatric disorders) | 1 (1)
Somnolence (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPM 962 (N=321)
Nausea (Gastrointestinal disorders) | 31 (38)
Dental Caries (Gastrointestinal disorders) | 20 (21)
Vomiting (Gastrointestinal disorders) | 16 (25)
Constipation (Gastrointestinal disorders) | 13 (13)
Stomatitis (Gastrointestinal disorders) | 8 (8)
Application Site Reaction (General disorders) | 198 (217)
Application Site Pruritus (General disorders) | 12 (13)
Oedema Peripheral (General disorders) | 12 (12)
Application Site Erythema (General disorders) | 10 (10)
Nasopharyngitis (Infections and infestations) | 76 (108)
Cystitis (Infections and infestations) | 11 (17)
Contusion (Injury, poisoning and procedural complications) | 24 (27)
Blood Creatine Phosphokinase Increased (Investigations) | 26 (27)
Weight Decreased (Investigations) | 8 (8)
Back Pain (Musculoskeletal and connective tissue disorders) | 20 (21)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (12)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 8 (8)
Dyskinesia (Nervous system disorders) | 50 (57)
Headache (Nervous system disorders) | 9 (14)
Posture Abnormal (Nervous system disorders) | 8 (8)
Hallucination Visual (Psychiatric disorders) | 34 (47)
Somnolence (Psychiatric disorders) | 21 (21)
Hallucination (Psychiatric disorders) | 16 (21)
Insomnia (Psychiatric disorders) | 7 (8)
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 11 (14)
Orthostatic Hypotension (Vascular disorders) | 15 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No